CLINICAL TRIAL: NCT05096507
Title: Perioperative Cytokines, Postoperative Delirium and Health Status in Older People Undergoing Hip Fracture Surgery - a Pilot Study
Brief Title: Cytokines, POD, Health Status, Older Hip Fracture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 21052
Record Dates: First submitted 2021-10-05; First posted 2021-10-27 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Postoperative Delirium; Hip Fracture Surgery; Older People
Keywords: Postoperative delirium; Older people; Cytokines; Self-reported Health Status
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample for Cytokine analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: People age 65 years and older undergoing primary hip fracture surgery
  Interventions: Procedure: Hip fracture Surgery (Primary)

INTERVENTIONS:
Procedure: Hip fracture Surgery (Primary) — Surgery for primary hip fracture requiring general or neuro-axial anaesthesia

SUMMARY:
An investigation of the change in inflammation marker levels across hip fracture surgery and an exploration of any association with change in self reported health status and incidence of postoperative delirium

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years old
* Admitted for primary hip fracture surgery

Exclusion Criteria:

* Preoperative cognitive impairment
* History of neurosurgery, neurologic diseases or head trauma
* Current systemic bacterial or viral infection
* Complex or multiple injuries

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients age ≥ 65 years old presenting to hospital with a primary hip fracture
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Cytokine dynamics | 2 days
  Difference preoperative serum cytokine levels and postoperative serum cytokine levels in pg/mL.
Incidence of postoperative delirium | 5 days
  Assessment for presence or absence of delirium during the post operative period.

SECONDARY OUTCOMES:
Self reported health related quality of Life | 120 days
  Assessed preoperatively and again at approximately 120 days after surgery using the EuroQol Five Dimension Five level (EQ-5D-5L) tool. The tool assesses on five aspects of health (Dimensions) and each dimension has five possible levels. The tool also has a visual analogue scale ranging from 0 (poorest) to 100 (best health)

CONTACTS AND LOCATIONS:
Overall Officials: Iain Moppett, DM, Principal Investigator — University of Nottingham
Locations (1):
- Queen's Medical Centre, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No